CLINICAL TRIAL: NCT04621240
Title: The BrainHealth Project - Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-32
Record Dates: First submitted 2020-04-28; First posted 2020-11-09 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online SMART Intervention & Stress Solutions (Experimental): Strategic Memory Advanced Reasoning Training (SMART) teaches meta-cognitive strategies for individuals to apply to their daily lives for improved performance
  Interventions: Behavioral: Online SMART & Stress Solutions

INTERVENTIONS:
Behavioral: Online SMART & Stress Solutions — 1. On-line SMART - (Strategic Memory Advanced Reasoning Training) is a curriculum that teaches strategies of how to use the brain better, in such a way that may improve brain health and performance. SMART strives to achieve optimal cognitive function realized by the brain's ability to efficiently manage complex information by abstracting its essential meaning rather than attempting to memorize details, and to prioritize the information in order to attend to the most relevant parts. 2. Stress Solutions - provides individuals with practical tools to enhance performance, reduce stress, build resilience and improve quality of life.

SUMMARY:
The proposed project is a pilot study in preparation for a larger study called The BrainHealth Project. The BrainHealth Project will be a prospective, longitudinal (10 yr) study focused on identifying determinants of brain health. Over the 4-month time commitment of this pilot study, 200 participants will complete online cognitive testing & functional magnetic resonance imaging (fMRI) at 2 time points (pre- and post-intervention). Up to 200 participants will complete online cognitive testing at 2 time points (pre- and post-intervention) and no fMRI. In between those time points, all participants will participate in online training and education regarding ways to optimize brain health, as well as overall health. Online training that will be recommended to participants include the following: (1) Strategic Memory Advanced Reasoning Training (SMART) teaches meta-cognitive strategies for individuals to apply to their daily lives for improved performance; and (2) Stress Solutions provides individuals with practical tools to reduce stress, build resilience and improve quality of life.

The main objectives are: (i) to characterize lifestyle, cognitive, and behavioral markers related to an individual's cognitive function from adolescent to elderly ages, (ii) to assess the neural/biological determinants predictive of maintenance of brain health, and (iii) to evaluate the impact of available cognitive and lifestyle interventions on improving and maintaining brain health.

DETAILED DESCRIPTION:
The Center for BrainHealth and Brain Performance Institute have years of experience working as a translational research facility with the mission of delivering evidence-based BrainHealth services to the public. However, as the goal of the larger project is to reach 120,000 individuals, this is only feasible through the use of online, remote interactions. Historically, the preponderance of experience at the Center for BrainHealth and Brain Performance Institute has been through face-to-face interactions. In order to make this shift to remote assessments, training, and interactions, we propose a pilot study of up to 400 healthy adults aimed at informing and perfecting the protocols for the larger study. In order to better understand any modifications or enhancements that may be required to the current online assessments and training, these pilot study participants will be selected from the local population, and will complete their BrainHealth Assessment, as well as complete online training.

The assessments and training included in this protocol consist of:

ASSESSMENTS

1. Online BrainHealth Index (2x) - a battery of measures of connected language, which have been found to be preserved in normal aging (see list of previous studies in the next section), combined with standardized neuropsychological measures that assess other areas of cognition such as attention, memory, visuospatial, executive and psychomotor functions.

   A. COGNITIVE (Recall. Learn. Solve. Innovate.) The COGNITIVE evaluation looks at how an individual thinks. We will look at complex thinking capacities - such as reasoning, flexibility, and strategy - and specific thinking components, such as processing speed, attention, and memory. (Completion time ~ 1 hour) BrainHealth Measures of Cognitive Performance - 30 minutes
   1. Strategic Memory: Visual Selective Learning Task
   2. Integrated Reasoning: Test of Strategic Learning (Test of Strategic Learning, TOSL part I)
   3. Innovation: Test of Strategic Learning (TOSL part II)
   4. Memory for Detail: Test of Strategic Learning (TOSL part III)

   Ace Measures of Cognitive Performance - 25 minutes
   1. Basic Response Time
   2. Color Blindness screening (non-editable)
   3. Visual Search, Top-Down Attention, Distraction Cost, Processing Cost
   4. Directed Attention
   5. Selective Attention, Interference Resolution
   6. Working Memory Updating Cognitive Flexibility

   B. EMOTIONAL Well Being (Mood. Centered. Perspective. Rebound.) The EMOTIONAL Well Being evaluation taps into an individual's emotional sense of yourself. We will ask how they feel about the quality of their life, their level of happiness, their levels of stress and sadness, and get a gauge on their emotional resilience. (Completion time: 15 min)
   1. Happiness: Oxford Happiness Questionnaire
   2. Life Satisfaction: Quality of Life Scale
   3. Resilience: Connor-Davidson Resilience Scale
   4. Depression, Anxiety, and Stress Scale (DASS-21)

   C. SOCIAL (Engage. Relate. Connect. Empathize.) The SOCIAL evaluation looks at an individual's social vibrancy and quality of relationships. We want to know how they feel about their social support networks and the meaningfulness of their social engagements. (Completion time: <8 min.)
   1. Amount of Positive Social Support: Social Support Survey Index
   2. Complexity of Social Interactions: Social BrainHealth Scale

   D. DAILY FUNCTION (Strive. Challenge. Habits. Responsibility.) The DAILY FUNCTION evaluation monitors the complexity (depth and breadth) of your daily responsibilities, habits, and challenges. We are interested in how you strive to optimize your life circumstances and habits.

   (Completion time: 20 minutes )
   1. Mindset: BrainHealth Appraisal Questionnaire
   2. Significance of Life Engagement: Engagement in Meaningful Activities Survey
   3. Sleep: Pittsburgh Sleep Quality Index
   4. Occupational Complexity: O*Net Database Census Coding
   5. Physical Exercise: Cardiorespiratory Fitness Estimate Questionnaire
2. Brain Imaging (2x)(resting state functional MRI), blood flow (Arterial Spin Labeling), cerebrovascular reactivity (CVR - with breath hold task) and white matter integrity (Diffusion MRI). In this pilot study, as well as the larger BrainHealth Project study, the neural data will be analyzed in conjunction with non-neural measures (cognitive, well-being, social engagement, sleep, etc.) to support the development of a reliable set of metrics to assess brain health.
3. Brain Gauge by Cortical Metrics (2x) - 15 minutes. The Brain Gauge is a cognitive assessment tool that measures brain health by testing sensory perceptions in the fingertips. This will be completed at the BrainPerformance Institute prior to imaging at the University of Texas (UT) Dallas BrainHealth Imaging Center. During each test, two orange tips on the Brain Gauge device will vibrate the pointer and middle finger on a participant's non-dominant hand in a specific way. The computer-based application will ask questions about what the participant felt. By measuring eight components of brain health (speed, focus, fatigue, accuracy, sequencing, timing perception, plasticity, and connectivity) the application will then analyze responses using clinically-proven neuroscience to provide a comprehensive mental fitness score called the CorticalMetric.

INTERVENTIONS Online Interventions 1. Strategic Memory Advanced Reasoning Training (SMART) is a curriculum that teaches strategies of how to use the brain better, in such a way that may improve brain health and performance. SMART strives to achieve optimal cognitive function realized by the brain's ability to efficiently manage complex information by abstracting its essential meaning rather than attempting to memorize details, and to prioritize the information in order to attend to the most relevant parts. Importantly, because this training is intended to improve cognition in the healthy population that is being studied in this submission, and is NOT treating or preventing a medical condition, it will not be classified as a medical device for the purposes of this study. Other similar online strategy-teaching curriculum in studies of healthy aging have set a precedent for this position, utilizing this rational.

2. Stress Solutions - provides individuals with practical tools to enhance performance, reduce stress, build resilience and improve quality of life. Training will include the neurophysiological effects of chronic stress and the neurophysiological impacts of mindfulness. Participants will learn and practice skills in awareness, self-regulation, and emotion regulation through attentional focus exercises grounded in mindfulness meditation. This training enables learners to recognize habitual, conditioned modes of reacting and resources the learner with skills to make a shift in their relationship to their thoughts, feelings and body sensations within conditions of chronic and acute distress.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18
* internet access and device
* fluent English speaker

Exclusion Criteria:

* Children are excluded from this study
* Individuals who do not speak or read English
* If individuals have undergone an in-person BrainHealth Index (previously BrainHealth Physical), they will need to wait 6 months have passed to participate.
* Individuals who will complete the imaging component must pass an fMRI screener and score a 26 or above on the TICS (Telephone Interview Cognitive Status)-M.
* A history of neurological disorders, injuries or disabilities (dementia, multiple sclerosis, Parkinson's, traumatic brain injury, stroke)
* A history of psychiatric disorders (schizophrenia, bipolar disorder, or others related to anxiety, depression, panic)
* A history of uncontrolled health issues (substance abuse, hypertension, hypo- or hyper-thyroidism)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Chapman, PhD, Principal Investigator — The Center for BrainHealth, University of Texas at Dallas
Locations (1):
- UTD Center for BrainHealth, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was all online and took place between March - Aug 2020
Pre-assignment Details: 200 participants were screened and 180 were enrolled
Period: Overall Study
Arm/Group | Online SMART Intervention & Stress Solutions
Started | 180
BrainHealth Index #1 | 180
Online Training | 174
BrainHealth Index #2 | 144
Completed | 144
Not Completed | 36
Not completed — Withdrawal by Subject | 36

BASELINE CHARACTERISTICS:
Arm/Group | Online SMART Intervention & Stress Solutions
Number analyzed (Participants) | 180
Age, Continuous [Mean (Full Range); unit: years] | 55.0 [18 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129
  Male | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic | 150
  Hispanic | 11
  Unknown | 19
Region of Enrollment [Number; unit: participants]
  United States | 180
BrainHealth Index [Median (Full Range); unit: units on a scale] | 54 [30 to 82]

OUTCOME MEASURES:

1. Primary Outcome: The BrainHealth Index
Description: The BrainHealth Index is a composite score of 22 individual measures encompassing four components of brain health, including (1) cognitive performance, (2) mental well-being, (3) daily life functioning (e.g., sleep, fitness, activities), and (4) social interactions/engagement. [Composite score min value = 30, Composite score max value = 82, higher composite score = better outcome]
Time Frame: 3 months
Population: Of the 180 generally healthy adults who completed their online baseline assessments, 144 completed their 3-month follow-up assessments.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Online SMART Intervention & Stress Solutions
Number analyzed (Participants) | 144
score on a scale | 54 [30 to 82]
Statistical Analysis 1: Comparison: Online SMART Intervention & Stress Solutions; Test type: Superiority — Mean level change from pre- to post-testing; p < 0.001, t-test, 2 sided; Mean Difference (Net) = 10.3
Statistical Analysis 2: Comparison: Online SMART Intervention & Stress Solutions; Test type: Other — Regression of the change in BrainHealth Index on age; p = 0.55, Regression, Linear; Slope = 0.03

ADVERSE EVENTS:
Time Frame: From day of enrollment (once participant passes screening and signs consent) to end of study (completion of second online assessment) (~3 months)
Description: Serious adverse events or death were not assessed, given the minimal risk nature of the study intervention and procedures
Arm/Group | Online SMART Intervention & Stress Solutions
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/180

LIMITATIONS AND CAVEATS:
Limitations include the following: (1) only one approach to cognitive training was examined in this study; others could be added for broader impact; (2) trainings and metrics around lifestyle factors will be enhanced with wearable technologies; (3) impact on broader cultural and socio-economic groups not well-understood; (4) not a randomized controlled trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT04621240/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT04621240/ICF_001.pdf